CLINICAL TRIAL: NCT02797509
Title: Preventing Chronic Depression and PTSD in Patients With Stroke Admitted to the Neuroscience ICU and Their Family Caregivers
Brief Title: Preventing Chronic Depression and PTSD in Stroke Patients Admitted to the Neuroscience Intensive Care Unit (NICU) and Their Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Ana-Maria Vranceanu, PhD, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P001190
Record Dates: First submitted 2016-06-02; First posted 2016-06-13 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Neurological Disorder
Keywords: Intensive Care Unit
MeSH Terms: conditions — Nervous System Diseases

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychosocial Skills-Based Intervention (Experimental): Based on information from Phase I (semi-structured interviews), the investigators will develop a detailed psychosocial intervention manual. The intervention will be tailored consistent with American Heart Association (AHA) recommendations for stroke skills based interventions and will include 2 general and 4 specific modules (selected from 7 available). Generally, in the intervention, stroke patients and stroke caregivers will learn skills to cope and manage stroke-related stressors. It is anticipated that the intervention will have 6 sessions with 2 general sessions delivered within the NICU face to face and 4 tailored specific sessions to be delivered via live video using Vidyo. Participants in the intervention group will also receive treatment as usual.
  Interventions: Behavioral: Psychosocial Skills-Based Intervention
- Minimally Enhanced Usual Care (MEUC) (No Intervention): Those in the MEUC will continue with their current care. This may include meeting with nurses, physical therapist, medical doctors, and other members of the stroke patient's medical team. Treatment as usual may also involve administration of Selective Serotonin Reuptake Inhibitors (SSRIs) to those patients with motor problems. They will also received a pamphlet with educational information on stroke and recovery

INTERVENTIONS:
Behavioral: Psychosocial Skills-Based Intervention — Subjects will attend group skills-based sessions once weekly (either in-person or via Vidyo) for 6 weeks and learn skills to cope and manage stroke-related stressors.
  Arms: Psychosocial Skills-Based Intervention

SUMMARY:
The current study has the following objectives:

1. To determine additional stroke patient (SP) and stroke caregiver (SC) factors including their perceptions of the stroke experience, hospitalization, and how they cope with its challenges; identify additional appropriate points to intervene (maladaptive coping styles, unrealistic expectations, inappropriate prioritization, misinformation about illness, and self care), and assess SP and SC preferences for the structure, mode of delivery (including potential for phone, video or a combination of these) and timing of an intervention.
2. To develop, [using the preliminary data and information from aim 1], and test the feasibility and acceptability (primary outcomes) of a skills-based intervention for preventing chronic depression, anxiety, PTSD and decreased QoL in dyads at risk.

ELIGIBILITY:
Eligible dyads (stroke patients and stroke caregivers) must meet the following inclusion criteria:

* Age 18 or older
* English fluency and literacy
* Hospitalized with an acute stroke (hemorrhagic and ischemic) within the past 2 weeks (patient) OR primary stroke caregiver of a stroke patient currently admitted with an acute stroke
* Stroke patient or stroke caregiver screens in for depression and/or PTSD

One or more of the following exclusion criteria will render a stroke patient (only) ineligible:

* Stroke patients who cannot participate due to the severity of stroke, cognitive impairment and/or aphasia, and are anticipated to not be able to participate due to permanent impairment as judged by the medical team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Feasibility of the Intervention | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Demonstration of feasibility will be assessed by the number of individuals who drop out of the study prior to completing the post- intervention assessment and the rate of missed sessions. If drop-out rate or missed-session rate exceeds 25%, revisions to the intervention may be needed.
Client Satisfaction Questionnaire (CSQ-8) | Change between post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Measures how satisfied the participant is with the intervention.

SECONDARY OUTCOMES:
Measure of Current Status (MOCS-A) | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Measures participants' current self-perceived status on several skills that are targeted by the intervention: the ability to relax at will, recognize stress-inducing situations, restructure maladaptive thoughts, be assertive about needs, and choose appropriate coping responses as needed.
Cognitive and Affective Mindfulness Scale (CAMS) | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Measures the degree to which individuals experience their thoughts and feelings.
World Health Organization QOL Questionnaire (WHOQOL-BREF) | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Measures one's perceptions in the context of their culture and value systems, and their personal goals, standards and concerns.
Modified Rankin Scale (mRS) | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Measures the patient's prior stroke status and stroke severity.
Hospital Anxiety and Depression Scale (HADS) | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Measures symptoms of anxiety and depression.
Posttraumatic Stress (PCL-S) | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Measures symptoms of posttraumatic stress disorder
Current psychotropic meds and comorbid medical conditions, | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Study staff will collect information on patient's medical history and current medications to measure their mental health throughout the study.
Barthel Index | Change between Baseline (week 0), post-intervention (week 8), 3-month Follow Up (week 13), and 6-month Follow Up (week 26)
  Measures the patient's prior stroke status and stroke severity.

OTHER OUTCOMES:
Age, Gender, Race, Ethnicity, Marital Status, Education Status, and Employment Status of Patients/Caregivers in the ICU | Baseline (week 0)
  This questionnaire asks ICU patients/caregivers to report their age, gender, race, ethnicity, marital status, highest level of education, and primary employment status over the last 12 months.
Credibility Questionnaire | Baseline (week 0)
  Measures how much the participant believes the intervention will work.
Prior Mental Health Questionnaire | Baseline (week 0)
  This questionnaire asks ICU patients/caregivers to report any previous or current mental health conditions that they have been diagnosed with in the past.

CONTACTS AND LOCATIONS:
Overall Officials: Ana-Maria Vranceanu, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bannon S, Lester EG, Gates MV, McCurley J, Lin A, Rosand J, Vranceanu AM. Recovering together: building resiliency in dyads of stroke patients and their caregivers at risk for chronic emotional distress; a feasibility study. Pilot Feasibility Stud. 2020 May 25;6:75. doi: 10.1186/s40814-020-00615-z. eCollection 2020. PMID 32509320